CLINICAL TRIAL: NCT05705024
Title: Efficacy of Locally Delivered Allogeneic Mesenchymal Stem Cells for Promoting Corneal Repair
Brief Title: Efficacy of Locally Delivered Allogeneic Mesenchymal Stromal Cells
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ali R Djalilian, Professor of Ophthalmology, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-0751; W81XWH-18-1-0661 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2023-01-21; First posted 2023-01-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Corneal Ulcer
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Thirty eight (38) patients will be recruited in this randomized clinical trial study with a 2:1 allocation for randomization. Twenty-five (25) patients will be recruited for the MSC treatment and thirteen (13) patients will be assigned to the control group. At any stage, if the results of MSC group were significantly better than the control group, using the control group would be stopped. This process will be supervised by Charlotte Joselin who is the person in charge for blinding and for the formulation and distribution of the proper study drug for injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Medium dose of allogenic MSC drops (Active Comparator): Dose of allogeneic MSC subconjunctival injection will be assigned 3,000,000 cells/150 µL.
  Interventions: Biological: Mesenchymal Stromal Cells
- Control Group (Sham Comparator): For the control group, 50 µL of the freezing media (vehicle) will be injected.
  Interventions: Other: Control Solution

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells — Subconjunctival Injection of Allogeneic Mesenchymal Stromal Cellsmasked clinical trial, patients with non-resolving corneal epithelial disease (i.e., refractory to standard treatments for at least two weeks) will receive a single subconjunctival injection of bone marrow-derived allogeneic MSCs or vehicle (CS5 freezing media, BioLife Solutions Inc, Bothell, WA, USA), with continued follow-up for up to 90 days.
  Arms: Medium dose of allogenic MSC drops
Other: Control Solution — For the control group, 150 µL of injectable normal saline (0.9% NaCl). will be injected.
  Arms: Control Group

SUMMARY:
The proposed Conventional Cohort Expansion Study involves the use of Mesenchymal Stromal Cells (MSCs) are derived from the bone marrow. We previously studied the safety of subconjunctival injection of allogeneic bone marrow-derived MSCs in patients with nonhealing epitheliopathy (IRB Protocol 2020-0334). In the present study, we want to study the efficacy of this treatment on chronic epitheliopathies.

DETAILED DESCRIPTION:
The "Efficacy of Locally Delivered Allogeneic Mesenchymal Stem Cells for Promoting Corneal Repair Study" otherwise known as the "MSC Study," is designed to assess the safety of allogeneic bone marrow-derived MSC secreted factor on the ocular surface via subconjunctival injection of MSC, and also obtain a preliminary observation on the following:

* Epithelial barrier integrity and/or wound closure.
* Development of Scarring.
* Final Visual Acuity.

The objective is to improve clinical outcomes in significant non-healing corneal wounds. To achieve these goals, the MSC Study will include a Phase II efficacy study.

ELIGIBILITY:
Inclusion Criteria:

Visual Acuity:

* Best corrected distance visual acuity (BCDVA) score ≤ 75 ETDRS letters, (≥ 0.2 LogMAR, ≤ 20/32 Snellen or ≤ 0.625 decimal fraction) in the affected eye.

Ocular Health:

* Patients with non-resolving corneal epitheliopathy or epithelial defect after two or more weeks of standard non-surgical treatments (e.g., preservative-free artificial tears, gels or ointments; discontinuation of preserved topical drops; anti-inflammatory therapy, soft bandage contact lens).
* No objective clinical evidence of improvement in the last 2 weeks (≤50% reduction in fluorescein staining or ≤50% reduction in longest diameter of the epithelial defect).
* If both eyes have chronic epithelial disease, the eye with the worse epithelial disease will be treated.
* Evidence of impaired epithelial barrier manifested by fluorescein staining of the epithelium with a score 10 or higher by National Eye Institute grading.
* Patients with stage 1 (no epithelial defect), stage 2 (persistent epithelial defect, PED; without stromal loss) or stage 3 (corneal ulcer; with stromal loss) neurotrophic keratopathy25-27 limited to ≤80% corneal diameter.

Study Procedures:

* Only patients who satisfy all Informed Consent requirements may be included in the study. The patient and/or his/her legal representative must read, sign and date the Informed Consent document before any study-related procedures are performed. The Informed Consent form signed by patients and/or legal representatives must have been approved by the IRB for the current study.
* Patients must have the ability and willingness to comply with study procedures.

Exclusion Criteria:

Visual Acuity:

* Best-corrected distance visual acuity (BCDVA) score better than 75 ETDRS letters, or 0.2 LogMAR, or 20/32 Snellen or 0.625 decimal fraction in the affected eye

Ocular Health:

* Ocular drug toxicity less than two weeks ago
* Any active ocular infection (bacterial, viral, fungal or protozoal) or active ocular inflammation in the affected eye.
* History of any ocular surgery (including laser or refractive surgical procedures) in the affected eye within the three months before study enrollment. (An exception to the preceding statement will be allowed if the ocular surgery is considered to be the cause of the PED. Ocular surgery in the affected eye will not be allowed during the study treatment period and elective ocular surgery procedures should not be planned during the duration of the follow-up period unless the patient will be involved in corneal thinning of more than 1/3 corneal stroma, corneal melting or perforation.
* Prior surgical procedure(s) for the treatment of a chronic corneal epitheliopathy (e.g., complete tarsorrhaphy, conjunctival flap, etc.) in the affected eye with the exception of amniotic membrane transplantation. Patients previously treated with amniotic membrane transplantation may only be enrolled two weeks after the membrane has disappeared within the area of the chronic corneal epitheliopathy or corneal ulcer or at least six weeks after the date of the amniotic membrane transplantation procedure. Patients previously treated with Botox (botulinum toxin) injections used to induce pharmacologic blepharoptosis are eligible for enrollment only if the last injection was given at least 90 days prior to enrollment in the study.
* Chronic corneal epitheliopathy in the background of endothelial decompensation that needs corneal graft
* Anticipated need for punctual occlusion during the study treatment period. Patients with punctual occlusion or punctual plugs inserted prior to the study are eligible for enrollment provided that the punctual occlusion is maintained during the study.
* Evidence of corneal ulceration involving the posterior third of the corneal stroma, corneal melting or perforation in the affected eye.
* Presence or history of any ocular or systemic disorder or condition that might hinder the efficacy of the study treatment or its evaluation, could possibly interfere with the interpretation of study results, or could be judged by the investigator to be incompatible with the study visit schedule or conduct (e.g., progressive or degenerative corneal or retinal conditions, uveitis, optic neuritis, poorly controlled diabetes, autoimmune disease, systemic infection, neoplastic diseases).
* Patients with uncontrolled eyelid abnormality that preclude appropriate eyelid closure or including eyelash abnormality

Study Procedures:

* Known hypersensitivity to one of the components of the study or procedural medications (e.g., fluorescein).
* History of drug, medication or alcohol abuse or addiction.
* Use of any investigational agent within 4 weeks of screening visit.
* Participation in another clinical study at the same time as the present study.
* Participants who are pregnant at the time of study enrollment will be excluded; pregnancy is identified according to the patient's self-report /positive βhCG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Improvement of Corneal Epithelial Barrier and/or Integrity (Efficacy Rate) | Day 28
  The proportion of patients with improved epithelial barrier and/or integrity from baseline to DAY 28 as determined by the investigator on slit lamp examination:
  * Improved epithelial barrier, defined as a 50 % improvement in corneal fluorescein staining score
  * Improved epithelial integrity, defined as a healed epithelial defect

SECONDARY OUTCOMES:
Visual Acuity | Baseline, Days 1-7, 28, 60, 90
  Percent change in best-corrected distance visual acuity from baseline to DAY 90, as measured using standard ETDRS protocols
Corneal staining and NEI grading | Baseline, Days 1-7, 28, 60, 90
  Grading of fluorescein staining of the cornea
Ocular Surface Parameters | Baseline, Day 28, 90
  Changes in tear breakup time (TBUT), ocular surface disease index (OSDI), Lissamine green staining, and anesthetic Schirmer's test from baseline to DAY 28 and DAY 90
Corneal Epithelial Thickness | Day 28, 90
  Percent change in corneal epithelial thickness from baseline to DAY 28 and DAY 90, as measured by anterior segment OCT (AS-OCT)
Patient Symptoms | Baseline, Days 1-7, 28, 60, 90
  Changes in ocular discomfort visual analog scale (VAS) 0 - 100, where 0 is no discomfort and 100 the worst discomfort, from baseline to DAY 90
Time to epithelial healing | Baseline, Days 1-7, 28, 60, 90
  Time of improvement of epitheliopathy
Corneal Scar | Baseline, Days 1-7, 28, 60, 90
  Change in the size of corneal scar (if present) from baseline to DAY 90, as documented by slit lamp photographs
Corneal Neo-vascularization | Baseline, Days 1-7, 28, 60, 90
  Change in corneal vascularization on slit lamp photographs from baseline to DAY 90
Conjunctival injection | Baseline, Days 1-7, 28, 60, 90
  Change in conjunctival injection on slit lamp examination from baseline to DAY 90

CONTACTS AND LOCATIONS:
Overall Officials: Ali R Djalilian, MD, Principal Investigator — University of Illinois at Chicago; Charlotte E Joslin, OD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (4):
- United States (4):
  - Department of Ophthalmology and Visual Sciences, Chicago, Illinois
  - University of Maryland at Baltimore, Baltimore, Maryland
  - Mass Eye and Ear Infirmary, Boston, Massachusetts
  - University of Pennsylvania, Scheie Eye Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cockerham GC, Lemke S, Rice TA, Wang G, Glynn-Milley C, Zumhagen L, Cockerham KP. Closed-globe injuries of the ocular surface associated with combat blast exposure. Ophthalmology. 2014 Nov;121(11):2165-72. doi: 10.1016/j.ophtha.2014.06.009. Epub 2014 Aug 11. PMID 25124272
- [Background] Cockerham GC, Lemke S, Glynn-Milley C, Zumhagen L, Cockerham KP. Visual performance and the ocular surface in traumatic brain injury. Ocul Surf. 2013 Jan;11(1):25-34. doi: 10.1016/j.jtos.2012.09.004. Epub 2012 Oct 5. PMID 23321357
- [Background] Cockerham GC, Rice TA, Hewes EH, Cockerham KP, Lemke S, Wang G, Lin RC, Glynn-Milley C, Zumhagen L. Closed-eye ocular injuries in the Iraq and Afghanistan wars. N Engl J Med. 2011 Jun 2;364(22):2172-3. doi: 10.1056/NEJMc1010683. No abstract available. PMID 21631351
- [Background] Baradaran-Rafii A, Eslani M, Tseng SC. Sulfur mustard-induced ocular surface disorders. Ocul Surf. 2011 Jul;9(3):163-78. doi: 10.1016/s1542-0124(11)70026-x. PMID 21791191
- [Background] Prockop DJ, Oh JY. Mesenchymal stem/stromal cells (MSCs): role as guardians of inflammation. Mol Ther. 2012 Jan;20(1):14-20. doi: 10.1038/mt.2011.211. Epub 2011 Oct 18. PMID 22008910
- [Background] Mittal SK, Omoto M, Amouzegar A, Sahu A, Rezazadeh A, Katikireddy KR, Shah DI, Sahu SK, Chauhan SK. Restoration of Corneal Transparency by Mesenchymal Stem Cells. Stem Cell Reports. 2016 Oct 11;7(4):583-590. doi: 10.1016/j.stemcr.2016.09.001. Epub 2016 Sep 29. PMID 27693426
- [Background] Wang LT, Ting CH, Yen ML, Liu KJ, Sytwu HK, Wu KK, Yen BL. Human mesenchymal stem cells (MSCs) for treatment towards immune- and inflammation-mediated diseases: review of current clinical trials. J Biomed Sci. 2016 Nov 4;23(1):76. doi: 10.1186/s12929-016-0289-5. PMID 27809910
- [Background] Yun YI, Park SY, Lee HJ, Ko JH, Kim MK, Wee WR, Reger RL, Gregory CA, Choi H, Fulcher SF, Prockop DJ, Oh JY. Comparison of the anti-inflammatory effects of induced pluripotent stem cell-derived and bone marrow-derived mesenchymal stromal cells in a murine model of corneal injury. Cytotherapy. 2017 Jan;19(1):28-35. doi: 10.1016/j.jcyt.2016.10.007. Epub 2016 Nov 10. PMID 27840134
- [Background] Ye J, Yao K, Kim JC. Mesenchymal stem cell transplantation in a rabbit corneal alkali burn model: engraftment and involvement in wound healing. Eye (Lond). 2006 Apr;20(4):482-90. doi: 10.1038/sj.eye.6701913. PMID 15895027
- [Background] Yao L, Li ZR, Su WR, Li YP, Lin ML, Zhang WX, Liu Y, Wan Q, Liang D. Role of mesenchymal stem cells on cornea wound healing induced by acute alkali burn. PLoS One. 2012;7(2):e30842. doi: 10.1371/journal.pone.0030842. Epub 2012 Feb 17. PMID 22363499
- [Background] Roddy GW, Oh JY, Lee RH, Bartosh TJ, Ylostalo J, Coble K, Rosa RH Jr, Prockop DJ. Action at a distance: systemically administered adult stem/progenitor cells (MSCs) reduce inflammatory damage to the cornea without engraftment and primarily by secretion of TNF-alpha stimulated gene/protein 6. Stem Cells. 2011 Oct;29(10):1572-9. doi: 10.1002/stem.708. PMID 21837654
- [Background] Oh JY, Kim MK, Shin MS, Lee HJ, Ko JH, Wee WR, Lee JH. The anti-inflammatory and anti-angiogenic role of mesenchymal stem cells in corneal wound healing following chemical injury. Stem Cells. 2008 Apr;26(4):1047-55. doi: 10.1634/stemcells.2007-0737. Epub 2008 Jan 10. PMID 18192235
- [Background] Ma Y, Xu Y, Xiao Z, Yang W, Zhang C, Song E, Du Y, Li L. Reconstruction of chemically burned rat corneal surface by bone marrow-derived human mesenchymal stem cells. Stem Cells. 2006 Feb;24(2):315-21. doi: 10.1634/stemcells.2005-0046. Epub 2005 Aug 18. PMID 16109757
- [Background] Li F, Zhao SZ. Control of Cross Talk between Angiogenesis and Inflammation by Mesenchymal Stem Cells for the Treatment of Ocular Surface Diseases. Stem Cells Int. 2016;2016:7961816. doi: 10.1155/2016/7961816. Epub 2016 Mar 24. PMID 27110252
- [Background] Cejkova J, Trosan P, Cejka C, Lencova A, Zajicova A, Javorkova E, Kubinova S, Sykova E, Holan V. Suppression of alkali-induced oxidative injury in the cornea by mesenchymal stem cells growing on nanofiber scaffolds and transferred onto the damaged corneal surface. Exp Eye Res. 2013 Nov;116:312-23. doi: 10.1016/j.exer.2013.10.002. Epub 2013 Oct 18. PMID 24145108
- [Background] Putra I, Shen X, Anwar KN, Rabiee B, Samaeekia R, Almazyad E, Giri P, Jabbehdari S, Hayat MR, Elhusseiny AM, Ghassemi M, Mahmud N, Edward DP, Joslin CE, Rosenblatt MI, Dana R, Eslani M, Hematti P, Djalilian AR. Preclinical Evaluation of the Safety and Efficacy of Cryopreserved Bone Marrow Mesenchymal Stromal Cells for Corneal Repair. Transl Vis Sci Technol. 2021 Aug 12;10(10):3. doi: 10.1167/tvst.10.10.3. PMID 34383879
- [Background] Jabbehdari S, Yazdanpanah G, Kanu LN, Anwar KN, Shen X, Rabiee B, Putra I, Eslani M, Rosenblatt MI, Hematti P, Djalilian AR. Reproducible Derivation and Expansion of Corneal Mesenchymal Stromal Cells for Therapeutic Applications. Transl Vis Sci Technol. 2020 Feb 21;9(3):26. doi: 10.1167/tvst.9.3.26. PMID 32742756
- [Background] Bartlett RS, Guille JT, Chen X, Christensen MB, Wang SF, Thibeault SL. Mesenchymal stromal cell injection promotes vocal fold scar repair without long-term engraftment. Cytotherapy. 2016 Oct;18(10):1284-96. doi: 10.1016/j.jcyt.2016.07.005. PMID 27637759
- [Background] Bara JJ, Richards RG, Alini M, Stoddart MJ. Concise review: Bone marrow-derived mesenchymal stem cells change phenotype following in vitro culture: implications for basic research and the clinic. Stem Cells. 2014 Jul;32(7):1713-23. doi: 10.1002/stem.1649. PMID 24449458
- [Background] Cook N, Hansen AR, Siu LL, Abdul Razak AR. Early phase clinical trials to identify optimal dosing and safety. Mol Oncol. 2015 May;9(5):997-1007. doi: 10.1016/j.molonc.2014.07.025. Epub 2014 Aug 14. PMID 25160636
- [Background] Al-Moujahed A, Chodosh J. Outcomes of an algorithmic approach to treating mild ocular alkali burns. JAMA Ophthalmol. 2015 Oct;133(10):1214-6. doi: 10.1001/jamaophthalmol.2015.2302. No abstract available. PMID 26226389
- [Background] Ghazaryan E, Zhang Y, He Y, Liu X, Li Y, Xie J, Su G. Mesenchymal stem cells in corneal neovascularization: Comparison of different application routes. Mol Med Rep. 2016 Oct;14(4):3104-12. doi: 10.3892/mmr.2016.5621. Epub 2016 Aug 11. PMID 27514011
- [Background] U.S. Department of Health and Human Services Food and Drug Administration Center for Biologics Evaluation and Research. Considerations for the Design of Early-Phase Clinical Trials of Cellular and Gene Therapy Products,. Accessed September 26, 2017. https://www.fda.gov/downloads/BiologicsBloodVaccines/GuidanceComplianceRegulatoryInformation/Guidances/CellularandGeneTherapy/UCM564952.pdf
- [Background] Sacchetti M, Lambiase A. Diagnosis and management of neurotrophic keratitis. Clin Ophthalmol. 2014 Mar 19;8:571-9. doi: 10.2147/OPTH.S45921. eCollection 2014. PMID 24672223
- [Background] Bonini S, Rama P, Olzi D, Lambiase A. Neurotrophic keratitis. Eye (Lond). 2003 Nov;17(8):989-95. doi: 10.1038/sj.eye.6700616. PMID 14631406
- [Background] Semeraro F, Forbice E, Romano V, Angi M, Romano MR, Filippelli ME, Di Iorio R, Costagliola C. Neurotrophic keratitis. Ophthalmologica. 2014;231(4):191-7. doi: 10.1159/000354380. Epub 2013 Oct 2. PMID 24107451
- [Background] Stevens S. Administering a subconjunctival injection. Community Eye Health. 2009 Mar;22(69):15. No abstract available. PMID 19506718
- [Background] Baradaran-Rafii A, Eslani M, Haq Z, Shirzadeh E, Huvard MJ, Djalilian AR. Current and Upcoming Therapies for Ocular Surface Chemical Injuries. Ocul Surf. 2017 Jan;15(1):48-64. doi: 10.1016/j.jtos.2016.09.002. Epub 2016 Sep 17. PMID 27650263
- [Background] Eslani M, Baradaran-Rafii A, Movahedan A, Djalilian AR. The ocular surface chemical burns. J Ophthalmol. 2014;2014:196827. doi: 10.1155/2014/196827. Epub 2014 Jul 1. PMID 25105018